CLINICAL TRIAL: NCT06096792
Title: Invastigation of the Relationship Between Early Quadriceps Arthrogenic Muscle Inhibition and Functional Recovery After Total Knee Arthroplasty
Brief Title: Muscle Recovery After Total Knee Arthroplasty
Status: Active, not recruiting | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Sibel Bozgeyik, Principal investigator, Hacettepe University
Other Study IDs: K-Bubble TKA
Record Dates: First submitted 2023-10-18; First posted 2023-10-24 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2024-10

CONDITIONS: Knee Arthritis, Osteoarthritis
Keywords: knee arthroplasty; Knee osteoarthritis; muscle inhibition
MeSH Terms: conditions — Osteoarthritis; Osteoarthritis, Knee

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Total knee arthroplasty (TKA) surgery is a common procedure performed to reduce pain, improve function, and enhance the quality of life in patients with end-stage knee osteoarthritis. As with other knee-related injuries and surgeries, TKA surgery can lead to inhibition of the quadriceps muscle, resulting in a decrease in the muscle's capacity to generate maximum voluntary force. This issue can negatively affect post-injury rehabilitation and function. The long-term persistent neuromuscular muscle inhibition in the quadriceps, one of the most important anti-gravity muscles in our body, leads to muscle atrophy and strength loss, which is more determinant in the development of functional limitations compared to joint range of motion and knee pain.

There have been no studies found that assess the quadriceps muscle inhibition occurring during the hospitalization of patients undergoing total knee arthroplasty surgery and examine its impact on post-discharge functional status.

The aim of this study is to evaluate the severity of arthrogenic inhibition in the quadriceps muscle of patients following total knee arthroplasty surgery, which is widely practiced in our country and considered the gold standard for the treatment of end-stage knee osteoarthritis. Additionally, the study aims to investigate its impact on post-discharge functional recovery. The data obtained from this study will provide guidance in monitoring patients' early functional recovery post-surgery and in better planning post-surgical rehabilitation.

The study will include patients aged 50-75 who have undergone total knee arthroplasty surgery due to knee osteoarthritis. Demographic information such as age, height, weight, and body mass index will be recorded. Pain will be assessed using a visual analog scale, and edema will be measured during hospitalization, at the 2nd and 6th-week follow-up visits. In addition to all the evaluations, functional status will be assessed at the 2nd and 6th-week follow-up visits using the 5-repetition sit-to-stand test, 10-meter walking test, and 2-minute walking tests, as well as knee function evaluated through the WOMAC and KOS-ADLS questionnaires.

DETAILED DESCRIPTION:
The study will include patients aged 50-75 who have undergone total knee arthroplasty surgery due to knee osteoarthritis. Demographic information such as age, height, weight, and body mass index will be recorded. Pain will be assessed using a visual analog scale, and edema will be measured during hospitalization, at the 2nd and 6th-week follow-up visits. In addition to all the evaluations, functional status will be assessed at the 2nd and 6th-week follow-up visits using the 5-repetition sit-to-stand test, 10-meter walking test, and 2-minute walking tests, as well as knee function evaluated through the WOMAC and KOS-ADLS questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Age between 50 and 75 years.
* Have undergone unilateral total knee arthroplasty surgery due to osteoarthritis.
* Hemodynamically stable post-surgery.
* Willing to participate in the study.

Exclusion Criteria:

* Having any neurological or oncological issues.
* Having undergone revision surgery.
* Having a history of cardiovascular surgery.

Ages: 50 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients who underwent total knee arthroplasty at Hacettepe University faculty of medicine
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2024-10-10 (Actual); Primary Completion 2025-03-20 (Actual); Study Completion 2025-09-11 (Estimated)

PRIMARY OUTCOMES:
muscle inhibition | postoperative day-1; postoperative day-2; postoperative day-3; postoperative 2th week and postoperative 6th week
  Quadriceps maximum isometric muscle contraction will be evaluated by measuring the pneumatic pressure change with a pneumatic dynamometer.

SECONDARY OUTCOMES:
Functional recovery | postoperative 2th week and postoperative 6th week
  Five times sit to stand test

CONTACTS AND LOCATIONS:
Overall Officials: Sibel Bozgeyik Bağdatlı, PhD, Principal Investigator — Hacettepe University
Locations (1):
- Hacettepe University, Ankara, Samanpazari, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided